CLINICAL TRIAL: NCT01144312
Title: Population Pharmacokinetics of Fentanyl in Patients Undergoing Living Donor Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Myung Hee Song/Assistant clinical professor, Department of Anesthesiology and Pain Medicine, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0534; 2009-0534 (Other: Asan Medical Center IRB)
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Living Donor Liver Transplantation
Keywords: LDLT
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pharmacokinetics of fentanyl (Experimental)
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — an initial intravenous bolus of fentanyl 100 μg and infusion of fentanyl at variable rates ranging from 250 to 400 μg/hr

SUMMARY:
The aim of this study was to characterize pharmacokinetics of fentanyl during and after Living Donor Liver Transplantation (LDLT), using population pharmacokinetic analysis with non linear mixed effects modeling.

DETAILED DESCRIPTION:
Patients received an initial intravenous bolus of fentanyl 100 μg and infused at variable rates ranging from 250 to 400 μg/hr.

Arterial blood samples (3ml) were taken immediately before the start of infusion (baseline), and at scheduled time which were coincident with laboratory tests during surgery as follows. In pre-anhepatic phase, blood were taken at 10min, 30min, 1hr, 3hr, 5hr until clamping of the hepatic blood supply and venous drainage, after the star of anhepatic phase, blood were taken at 5 min, 10 min, 30 min, 60 min, 90 min, 2hr until the vessels were reconnected to new liver. In neo-hepatic phase, blood were taken at 5min, 10min, 30min, 60min, 90min, 2hr, 3hr, 5hr until fentanyl-infusion stop, and at 0hr, 1hr, 3hr, 5hr, 8hr, 12hr, 24hr immediately after the stop of infusion. Samples were collected into tubes containing heparin as an anticoagulant and immediately placed on ice. After centrifugation for 8 min at 1800 g, the plasma was transferred to a cryovial and stored at -70°C until assay.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 19 - 65 years of age
* Over 45kg of weight
* Written Informed consent
* Patients receiving a liver graft from living donor (ASA PS III or IV)

Exclusion Criteria:

* Patients with renal dysfunction
* Patients with Fulminant hepatic failure
* Patients participated other clinical trials within 2 months
* Unable or Unwilling to give informed consent
* Abnormal test results with clinical significance

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters of fentanyl during LDLT | 48 Hours (during anesthesia of LT and after infusion stop)
  characterize pharmacokinetics of fentanyl during and after LDLT, using population pharmacokinetic analysis with non-linear mixed effects modeling.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea